CLINICAL TRIAL: NCT00807339
Title: CyberKnife Stereotactic Radiation for Unresectable Renal Tumors/PhaseI Study
Brief Title: CyberKnife for Unresectable Renal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Irving Kaplan, Assistant Professor of Radiation Oncology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005P00384
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Renal Cancer
Keywords: CyberKnife
MeSH Terms: conditions — Kidney Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Phase I dose escalation
  Interventions: Radiation: Stereotactic radiation; Device: CyberKnife Robotic Radiosurgery System

INTERVENTIONS:
Radiation: Stereotactic radiation — Dose escalation three consecutive treatments
Device: CyberKnife Robotic Radiosurgery System

SUMMARY:
This is a dose escalation study using the CyberKnife radiotherapy device for small surgical or medically untreatable renal tumors. Patients with renal tumors 5cms or less in diameter will be accrued onto this study. The ability of CyberKnife to ablate these renal tumors and maintain renal function with dose escalation will be assessed.

DETAILED DESCRIPTION:
The CyberKnife Robotic Radiosurgery System is a unique radiosurgical system capable of treating tumors anywhere in the body noninvasively and with sub-millimeter accuracy. The CyberKnife System delivers radiation using a precise targeting methodology allowing a focal treatment margin around the target, thus limiting the volume of adjacent tissue receiving high doses radiation. This in turn allows the delivery of high doses of radiation to the prostate over a short series of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Tumor size 5 cm or less
* Radiographic evidence of malignancy or Histologically verified primary renal malignancy.
* If the kidney biopsy is inconclusive but the radiologist determines that the tumor based on the CT/MRI is highly suspicious for cancer, you may participate
* Patients with highly suspicious lesions on CT or MRI
* One -three gold fiducials placed in or around tumor
* Contradiction or patient refusal to partial or complete nephrectomy
* Age 18 or greater
* KPS score 70 or greater

Exclusion Criteria:

* Irreversible coagulopathies that preclude fiducial placement

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2014-08-20 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of CyberKnife radiation | 2 years

SECONDARY OUTCOMES:
To evaluate local control, overall survival and late toxicity including preservation of renal function | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No